CLINICAL TRIAL: NCT01926210
Title: The Comparison of Mild Stimulation and Controlled Ovarian Stimulation in Poor Ovarian Responders: a Prospective Randomized Study.
Brief Title: Comparison of Ovarian Mild Stimulation and Controlled Ovarian Stimulation in Poor Ovarian Responders
Acronym: POR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Huang Rui (Other)
Responsible Party: Sponsor-Investigator, Huang Rui, M.D., Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A-2013-01-05S
Record Dates: First submitted 2013-08-14; First posted 2013-08-20 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2013-08

CONDITIONS: Infertility
Keywords: Poor ovarian response; in vitro fertilization; mild ovarian stimulation; controlled ovarian stimulation
MeSH Terms: conditions — Infertility | interventions — Letrozole; LHRH, Ac-Nal(1)-Cpa(2)-Trp(3)-Arg(6)-Ala(10)-; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mild ovarian stimulation (Experimental): Patients are stimulated with mild ovarian stimulation protocol,i.ed, from cycle day 3 to 7, letrozole 5mg per day are administrated and recombinant FSH 150 IU are given on day 4 and 6 . On cycle day 8, serum FSH LH, and estradiol levels are measured, and after then, the dose of recombinant FSH is adjusted according to the ovarian response and the maxim recombinant FSH dose is 150 IU/d. The GnRH-antagonist (Cetrotide) 0.25mg per day is administrated when the estradiol level reaches 200 pg/ml and the serum LH level rises above 2 times of basal LH level.
  Interventions: Other: mild stimulation protocol
- controlled ovarian stimulation (Active Comparator): Patients are stimulated using controlled ovarian stimulation protocol,i.e., from cycle day 18-22 (day 7 after ovulation) of previous cycle, all participants are given short-acting GnRH agonist (Triptorelin 0.05mg/d) for 14 days, then after checking serum FSH, LH and estradiol to make sure that complete downregulation is achieved, exogenous gonadotropin (recombinant FSH) 300 IU/d is given for 5 days, then the dose of recombinant FSH is adjusted according to ovarian response.
  Interventions: Other: controlled ovarian stimulation

INTERVENTIONS:
Other: mild stimulation protocol — letrozole is used from cycle day 3 to 7 and low dose recombinant FSH(no more than 150 IU/d) is used on cycle day 4,6 and 8 onwards. GnRH antagonist is only applied in case of premature LH rise might happen.
  Other Names: letrozole; recombinant FSH; GnRH antagonist
  Arms: mild ovarian stimulation
Other: controlled ovarian stimulation — After fully downregulation by using short-acting GnRH agonist, 300 IU/d recombinant FSH is administrated for 5 days, then the dose is adjusted according to ovarian response.
  Other Names: GnRH agonist; recombinant FSH
  Arms: controlled ovarian stimulation

SUMMARY:
This is a prospective, randomized clinical trial to compare the efficiency and safety of mild stimulation and controlled ovarian stimulation protocol on the treatment of POR. The randomization is achieved on the basis of a computer-generated randomization list in a 1:1 ratio.

DETAILED DESCRIPTION:
500 poor ovarian responders will be equally randomized to two different ovarian stimulation protocol arms,i.e, mild ovarian stimulation(experimental arm) or controlled ovarian stimulation(control arm). In experimental arm, patients will received letrozole 5mg per day from cycle day 3 to 7 and recombinant follicle-stimulating hormone (FSH) 150 international unit (IU) on day 4 and 6. The dose of recombinant FSH is adjusted according to the ovarian response and the gonadotropin-releasing hormone(GnRH)antagonist(Cetrotide) 0.25mg per day is administrated when the estradiol level reaches 200 pg/ml and the serum luteinizing hormone （LH）level rises above 2 times of basal LH level. In control arm,patients will be stimulated with short-acting GnRH agonist long protocol. After complete downregulation is achieved through GnRH-agonist, recombinant FSH 300 IU/d is given for 5 days, then the dose of recombinant FSH is adjusted according to ovarian response.

The clinical and ongoing pregnancy rate and other secondary outcome parameters are compared between these two groups.

ELIGIBILITY:
Inclusion Criteria:

* a. Poor ovarian responders b. Normal BMI (18-25 Kg/m2) c. Regular menstruation (with cycle 23-35 days)

Exclusion Criteria:

* a. History of repeated IVF failure (previous IVF cycle >2) b. Serious adenomyosis c. Polycystic ovary syndrome(PCOS) patients d. History of allergic to ovulation induction medicines e. Abnormal uterine cavity, i.e, intrauterine adhesion f. Attending other clinical trials in the same period. g. History of systemic disease contradictory to COH or pregnancy.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy rate | 7 weeks

SECONDARY OUTCOMES:
live birth rate | 10 months
Number of oocytes retrieved | 3 weeks
Number of transferrable embryo | 3 weeks
normal fertilization rate | 3 weeks
implantation rate | 7 weeks
ongoing pregnancy rate | 3 months
Total dose of recombinant FSH consumption | 3 weeks
length of stimulation | 3 weeks
serum estradiol level | 3 weeks
serum LH level | 3 weeks
serum progesterone level | 3 weeks
serum FSH level | 3 weeks
FSH level in follicular fluid | 3 weeks
LH level in follicular fluid | 3 weeks
Estradiol level in the follicular fluid | 3 weeks
progesterone level in follicular fluid | 3 weeks
testerone level in the follicular fluid | 3 weeks
anti-müllerian hormone (AMH)level in follicular fluid | 3 weeks
Ovarian Hyperstimulation Syndrome (OHSS) rate | 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rui Huang, M.D., Principal Investigator — sixth affiliated hospital of Sun Yet-san University
Locations (1):
- sixth affiliated hospital of Sun Yet-san University, Guangzhou, Guangdong, China